CLINICAL TRIAL: NCT01420913
Title: Randomized,Open-label,Parallel Study to Evaluate the Pharmacokinetic Characteristics of Pregabalin According to Different Controlled Released Formulations in Healthy Male Subjects
Brief Title: Randomized, Open-label, Parallel Study to Evaluate the Pharmacokinetic Characteristics of Pregabalin According to Different Controlled Released Formulations in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: YCD207
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: To evaluate the pharmacokinetic characteristics of Lyrica, YHD1119 A,B,C
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lyrica capsule(Pregabalin 150mg) (Active Comparator)
  Interventions: Drug: Pregabalin
- YHD1119 A(Pregabalin SR 300mg) (Experimental)
  Interventions: Drug: Pregabalin
- YHD1119 B(Pregabalin SR 300mg) (Experimental)
  Interventions: Drug: Pregabalin
- YHD1119 C(Pregabalin SR 300mg) (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 300mg a day

SUMMARY:
The purpose of this trial is to compare the pharmacokinetic characteristics of YHD1119 A, YHD1119 B, YHD1119 C and Lyrica capsule.

YHD1119 A, B, C are controlled released formulations which are made by YUHAN Corporation.

Primary endpoints are C max,ss and AUC tau. Secondary endpoints are AUC last, AUC infinity, T max,ss, t 1/2

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, healthy adult male subject
* >55 Kg(Body weight) and < ideal body weight ± 20%

Exclusion Criteria:

* AST or ALT > 1.25 * Upper normal range (Lab)
* Total bilirubin > 1.5 * Upper normal range
* Systolic BP >140 OR <100, Diastolic BP >90 OR <65

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | 36 hr
AUCtau | 36 hr
Safety monitoring | 14 days
  Laboratory findings Adverse event

SECONDARY OUTCOMES:
AUClast AUCinfinity Tmax,ss t1/2 | 36 hour
AUCinfinity | 36 hr
Tmax,ss | 36 hr
t 1/2 | 36 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul ST.Mary Hospital, Seoul, South Korea